CLINICAL TRIAL: NCT05279326
Title: Virtual Shared Medical Appointments (SMAs) in Lifestyle Approach for Type 2 Diabetes: Protocol of a Randomized Pragmatic Trial
Brief Title: Virtual SMAs in Lifestyle Approach for Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Unidade de Saúde Familiar Homem do Leme (Unknown); Health4All Primary Healthcare Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMAs
Record Dates: First submitted 2022-02-14; First posted 2022-03-15 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants will receive virtual SMAs and usual care. Virtual SMAs will last 90 minutes, every 3 weeks, in 18 weeks through an online platform, at no cost to participants beyond the use of the device and the internet.
  Interventions: Behavioral: Virtual SMAs
- Control arm (No Intervention): Participants will be at usual care and follow their usual contact with health services.

INTERVENTIONS:
Behavioral: Virtual SMAs — 18 weeks lifestyle approach for type 2 diabetes program: Session 1 (week 0): Introduction; Session 2 (week 3): Behaviour change process; Session 3 (week 6): Medical nutrition therapy recommendations - Part 1; Session 4 (week 9): Medical nutrition therapy recommendations - Part 2; Session 5 (week 12): Medical physical Activity recommendations; Session 6 (week 15): Smoking cessation: tobacco and E-cigarettes; Session 7 (week 18): Diabetes distress.
  Arms: Intervention arm

SUMMARY:
This study protocol presents the design of a randomized pragmatic trial. This study aims to determine the effectiveness of virtual shared medical appointments (SMAs) lifestyle approach in improving glycaemic control, compared to usual care in type 2 diabetes (T2D) subjects.

ELIGIBILITY:
Inclusion Criteria:

* (1) be 18 years old or older
* (2) have a diagnosis of T2D with HbA1c ≥ 6.5% within the preceding 6 months
* (3) have body mass index (BMI) ≥ 25.0 kg/m2 within the preceding 6 months
* (4) have access to a camera and internet

Exclusion Criteria:

* unable to attend virtual SMAs for diagnosis of dementia or other cognitive impairment and any behavioral problem, which interferes with group participation and discussion
* not fluent in Portuguese, and unable to follow conversations, read instructions, and read in Portuguese
* being pregnant or planning a pregnancy in the next year
* attending a weight loss and/or physical activity counseling program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in glycaemic management, to be assessed by blood analysis | 12 months
  Difference between the intervention and control group in the change of serum glycated hemoglobin A1c (HbA1c) concentrations from baseline to the end of follow-up.

SECONDARY OUTCOMES:
Change in weight, to be assessed by weight balance | 12 months
  Difference between the intervention and control group in the change of weight from baseline to the end of follow-up.
Change in waist circumference, to be assessed by measuring tape | 12 months
  Difference between the intervention and control group in the change of waist circumference from baseline to the end of follow-up.
Change in systolic and diastolic blood pressure, to be assessed by sphygmomanometer | 12 months
  Difference between the intervention and control group in the change in systolic and diastolic blood pressure from baseline to the end of follow-up.
Change in fasting plasma triglycerides concentrations, to be assessed by blood analysis | 12 months
  Difference between the intervention and control group in the change of serum triglycerides concentrations from baseline to the end of follow-up.
Change in fasting plasma low density lipoprotein (LDL) concentrations, to be assessed by blood analysis | 12 months
  Difference between the intervention and control group in the change of serum low density lipoprotein (LDL) concentrations from baseline to the end of follow-up.
Change in fasting plasma high density lipoprotein (HDL) concentrations, to be assessed by blood analysis | 12 months
  Difference between the intervention and control group in the change of serum high density lipoprotein (HDL) concentrations from baseline to the end of follow-up.
Change in number of individual consultations, to be assessed by electronic health record | 12 months
  Difference between the intervention and control group in the change of number of individual consultations from baseline to the end of follow-up.
Change in use of medication, to be assessed by electronic health record | 12 months
  Difference between the intervention and control group in the change of the use of medication from baseline to the end of follow-up.
Change in the participants' satisfaction, to be assessed by questionnaire | 12 months
  Difference between the intervention and control group in the participants' satisfaction from baseline to the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalia Pascoa, MD, PhDc, Principal Investigator — Universidade do Porto
Locations (1):
- Unidade de Saúde Familiar Homem do Leme, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No